CLINICAL TRIAL: NCT04470960
Title: Evaluation of a Health Promoting Community Center Network (HPCCN) Innovation
Acronym: HPCCN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Ministry of Health, Israel (Other Government)
Responsible Party: Principal Investigator, Donna R Zwas, Director of The Linda Joy Pollin Womens Cardiovascular wellness Center, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ccproject-HMO-CTIL
Record Dates: First submitted 2020-03-01; First posted 2020-07-14 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: A Community Center as a Health Promoting Setting
Keywords: Community Centre; Healthy setting; Health promotion; framework formation

STUDY DESIGN:
Intervention Model Description: A framework is being evaluated in order to assess if a Community center has the capacity of serving as a healthy setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participating community centers (Experimental): Training course for the community center health coordinators Professional guidance for the CC health coordinators
  Interventions: Behavioral: Training course for the community center health coordinators

INTERVENTIONS:
Behavioral: Training course for the community center health coordinators — These community centers who have volunteered to join the project will receive a 12 week training session which includes the values and principles of health promotion and the principles of building a health promotion project.
  The participants will be requested to build a health promotion project within their community. Building and implementing the project will be assisted by a health promotion specialist. Each health promotion project will be evaluated according to the principles of health promotion.
  Other Names: Professional guidance for the CC health coordinators

SUMMARY:
The purpose of this research study is to design, implement and evaluate the setting for a "Healthy Community Center". This is a program review of a program which will be planned in a community based participatory level, based on the socioecological model. A pre-post design will be utilized where all community centers in the study will be exposed to the intervention components. It is hypothesized that community centers who will receive the intervention will have better skills at building sustainable participatory effective health promotion projects and will provide a healthy setting for the community within its juristiction.

DETAILED DESCRIPTION:
The purpose of this research study is to design, implement and evaluate the setting for a "Healthy Community Center". This is a program review of a program which will be planned in a community based participatory level, based on the socioecological model. A pre-post design will be utilized where all community centers in the study will be exposed to the intervention components. All community centers (n=15) will be evaluated by pre intervention questionairres and focus groups of community center Managers and health promotion professionals. The network will be designed upon the foundation of the "Healthy Cities network" with adaptations made in the process of participatory planning and designing according to the results of the focus groups. Intervention will include a a 12 week training session for designated "Health Coordinator" from each community center, Planning and implementing a personolized Health promtion Project in each community centre .It is hypothesized that community centers who will receive the intervention will have better skills at building sustainable participatory effective health promotion projects and will provide a healthy setting for the community within its juristiction.

ELIGIBILITY:
Inclusion Criteria:

* People who live within the geographical area of the community centers

Exclusion Criteria:

* Children under the age of 6 People who do not reside within the geographical area of the community centers

Min Age: 6 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
project planning, implementation and assessment | 3 years
  RE-AIM assessment of Reach, Effectiveness, Adoption, Implementation and Maintenance of the Community Center Programs, assessed by interview, There are 4-6 tailored questions in each domain and the answers are coded as yes, partially and no. Scores range from 0 -93
Israeli Healthy Cities Network adapted measure | 12 months after intervention initiation
  Israeli Healthy Cities Network evaluation tool was designed based on the MARI's (Monitoring Accountability Reporting Impact assessment) framework. It assesses six dimensions of the principles and strategies of the Healthy Cities work: (i) Equity policy and political support. (ii) Management. (iii) Health promotion programs and activities in the city. (iv) Community participation. (v) Intersectoral partnerships (vi) Environmental protection activities. This questionnaire was adapted to a community center framework.

SECONDARY OUTCOMES:
European Quality Instrument for Health Promotion | 6 months after intervention initiation
  information on four domains using in-person interviews: (i) compliance with international principles of Health promotion programs, (ii) development and implementation, (iii) project management and (iv) sustainability of programs. each item of the EQUIHP tool was recoded on a scale of 0-1: a score of 0 if the criteria was identified as not fulfilled, 0.5 if partly fulfilled and 1 if fully fulfilled. The sum of all valid scores per programme was divided by the number of valid answers to give the mean score. A mean score was given for each of the four domains, and for the overall score in the same manner. Higher scores are better.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Derived] Barasche-Berdah D, Wetzler S, Greenshtein I, Greenberg KL, Leiter E, Donchin M, Zwas DR. Municipal community centers as healthy settings: evaluation of a real-world health promotion intervention in Jerusalem. BMC Public Health. 2022 Oct 7;22(1):1870. doi: 10.1186/s12889-022-14220-7. PMID 36207706